CLINICAL TRIAL: NCT06242613
Title: National Multicenter Cohort Study of Robot-Assisted Gastrectomy Versus Laparoscopy in Gastric Cancer
Acronym: ROBOTAG
Status: Enrolling by invitation | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, MARÍA ASUNCIÓN ACOSTA MÉRIDA, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: ROBOTAG
Record Dates: First submitted 2023-01-18; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
Keywords: Gastrectomy; Lymphadenectomy; Robotic Surgery; Laparoscopic Surgery; Robot Assisted Gastrectomy; Laparoscopic Gastrectomy; Gastric Surgery; Minimally Invasive Gastrectomy; Robotic Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic Surgery: Patients underwent gastric surgery through the use of a robotic system.
  Interventions: Procedure: Robot-Assisted Gastrectomy
- Laparoscopic Surgery: Patients underwent gastric surgery with laparoscopic procedures.
  Interventions: Procedure: Laparoscopic Gastrectomy

INTERVENTIONS:
Procedure: Robot-Assisted Gastrectomy — Gastrectomy performed with a robotic system.
  Groups: Robotic Surgery
Procedure: Laparoscopic Gastrectomy — Gastrectomy performed with conventional laparoscopic approach.
  Groups: Laparoscopic Surgery

SUMMARY:
In recent years there has been a rapid incursion of robotic technology applied to almost all fields of surgery. In gastric cancer, whose mainstay of treatment is still surgical resection, gastrectomy with robotic lymphadenectomy is growing faster than the scientific evidence supporting its results.

The "National Multicenter Cohort Study of ROBOT-Assisted Gastrectomy Versus Laparoscopy in Gastric Cancer" (ROBOTAG study) is proposed as a prospective multicenter Spanish nationwide study, comparing robotic gastrectomy versus conventional laparoscopic gastrectomy for the treatment of gastric cancer. This study aims to provide evidence on the feasibility, safety and complications, possible technical advantages, short and long term surgical and oncological results, as well as aspects related to quality of life, which can support the increase in cost and the important technological effort that underlies robotic surgery with respect to conventional laparoscopic access.

The relevance of this project is doubled by directing the objectives, on the one hand, on a new and expensive technology that is reaching hospitals still surrounded by controversy about its real benefits; and on the other hand, by acting on a pathology for which most of the available studies come from Eastern countries, sometimes not very applicable to the Western context.

DETAILED DESCRIPTION:
RELEVANCE OF THE STUDY

The project presented here is a pioneering study in Spain, which aims to provide scientific evidence on robot-assisted gastrectomy in gastric cancer. The feasibility, oncologic outcomes, potential benefits, complications and limitations will be investigated. Few hospitals in the country have robotic technology and also perform this surgical procedure. The aim is to include as many centers as possible in this study, which will involve an important effort, but also the search for answers of great scientific value and repercussion in the applicability of this innovation in western environment. It is hoped to be able to provide, both at the management level of the Spanish Health System and extensively in other countries, a basis for decision making to audit and, if necessary, endorse the development and diffusion of this technology in hospitals, in order to offer patients the best surgical option in the treatment of gastric cancer.

OBJECTIVES

The main objective of this study is to compare Robot-Assisted Gastrectomy (RAG) with conventional Laparoscopic Gastrectomy (LG), from the point of view of clinical and oncological safety.

In addition, possible differences between patients undergoing each technique will be analyzed in other aspects, both intraoperatively and postoperatively.

Primary objective The main objective of this study is to compare the clinical and oncological safety of robot-assisted gastrectomy (RAG) with conventional laparoscopic gastrectomy (LG).

For this purpose the investigators will analyze in both groups (robot and laparoscopy):

1. as a measure of clinical safety:

   * Intraoperative blood loss
   * Perioperative complications
2. and as a measure of oncologic safety:

   * Nodal count (Number of lymph nodes retrieved)
   * R0 resection margin

   Secondary objectives

   To assess the differences between the groups (RAG vs LG) in intraoperative outcomes:
   * Operative time
   * Number of surgeons per procedure
   * Need for conversion to open surgery
   * Surgeon comfort
   * Learning curve

   To assess the differences between groups (RAG vs LG) in postoperative recovery course and physical status:
   * Onset of oral tolerance
   * Onset of mobilization
   * Hospital stay
   * Readmission
   * Mortality.

   To assess the differences between groups (RAG vs LG) in oncological outcomes:
   * Overall and disease-free survival
   * Local and systemic recurrence To assess the differences between the groups (RAG vs LG) cost utility measured in QALYs.

   HYPOTHESIS

   Robot-assisted laparoscopic gastrectomy with lymphadenectomy (RAG) offers at least the same results as gastrectomy with lymphadenectomy using a conventional laparoscopic (LG) approach in the treatment of gastric cancer, in terms of feasibility, safety, complications, and oncological outcomes.

   MATERIAL AND METHODS
   * Type of study: National, multicenter, prospective follow-up cohort study in patients undergoing minimally invasive gastric cancer surgery, using robot-assisted laparoscopic gastrectomy with lymphadenectomy (RAG) versus conventional laparoscopy (LG).
   * Study population: Patients diagnosed with gastric adenocarcinoma, in whom surgical treatment with curative intent by minimally invasive gastrectomy (RAG or LG) has been indicated.

   The protocol will follow standard clinical practice, without being modified by the present study.

   Patients who agree to participate in the study will have signed the informed consent form.

   • Primary outcome variable:
   * As a clinical safety measure, intraoperative blood loss and perioperative complications at 30 and 90 days will be analyzed.
   * As an oncological safety measure, the number of resected lymph nodes and the R0 resection margin will be analyzed.
   * Other intraoperative and postoperative, oncologic and quality of life parameters will be analyzed secondarily.

     * Sample size:

   This study aims to involve the largest number of centers nationwide and recruit the largest possible number of patients that these centers can provide. Taking into account the annual incidence of cases in each center, an approximate number of 20 cases per year per center is estimated. With the participation of at least 20 hospital centers, the investigators hope to obtain a sample of at least 400 patients for analysis.
   * Inclusion criteria:

     - Histologically confirmed primary gastric adenocarcinoma

     - Clinical stages Ib, II and III of gastric cancer (8th edition of the TNM classification)

     - Patients with ECOG performance status 0, 1 or 2

     - Patients who sign the informed consent to participate in the study

     - Patients over 18 years old

     - Patients treated by surgery with curative intent
   * Exclusion criteria:

     - Any histology other than adenocarcinoma

     - Stage Ia and IV

     - Unresectability criteria (tumor factors): distant metastasis, peritoneal carcinomatosis, positive cytology of ascitic fluid, invasion or tumor entrapment of large vessels (aorta, liver, celiac trunk), infiltration of the root of the mesentery, para-aortic lymphadenopathy or levels >3, linitis plastica, involvement of other organs

     - Inoperability criteria (patient factors): serious concomitant systemic disorders incompatible with surgery or the study (at the discretion of the investigator)

     - Non-compliance with any of the inclusion criteria
     * Patients undergoing surgery for gastric cancer with open approach at the beginning
     * Palliative surgery cases
   * Recruitment:

   All the centers included in the study must have the human and technical means necessary to guarantee the quality of the surgical treatment of gastric cancer, following current standards.

   The surgery will be performed in a hospital that has a specialized Esophagogastric Surgery Unit that performs advanced minimally invasive, laparoscopic and robotic surgery on a regular basis, as well as a Multidisciplinary Tumor Committee.

   All surgeons included must have previous experience of at least 20 gastrectomies with laparoscopic lymphadenectomies and an annual caseload of at least 10 cases; in addition to having accreditation as a robot console surgeon, having previously performed at least 3 gastrectomies with robot-assisted oncologic lymphadenectomy.

   Patients who are candidates for inclusion by the participating centers, who meet the inclusion criteria and who wish to participate, must sign the informed consent for the study. Access codes will be assigned to the center's investigators for the anonymized introduction of the study data. The confidentiality of the information handling of this study will be guaranteed, following national and international regulations.

   • Duration of study: Each collaborating researcher will provide patients who meet the inclusion criteria, recruiting them for 1 year. The minimum follow-up of all patients will be 1 year, after which the global analysis of the data and the corresponding study will be carried out. The final objective would be to achieve follow-up of all patients for at least 5 years, after which a new global analysis of the sample would be carried out to obtain the results after this period.

   • Follow-up: All patients included in the study must have at least a 1-year follow-up.

   The study will end when all enrolled patients have been followed for five years, died, withdrew consent or were lost to follow-up. A preliminary analysis of results will be performed when all patients enrolled in the study have been followed for the first year.

   • Data collection:

   In this study it is planned to obtain information from the collection of preoperative, intraoperative and postoperative data:

   - Patient's affiliation data

   - Medical history

   - Analytical and complementary test data

   - Patient and tumor characteristics

   - Surgical procedure parameters
   * Postoperative results
   * Follow-up data and quality of life

   The patient will be followed up throughout the study, and the status of the postoperative variables will be collected at each medical appointment.

   • Statistical analysis: Descriptive analysis of the data will be performed. Qualitative variables will be presented by frequency distribution and quantitative variables will be measured by indicators of central tendency (mean or median) and dispersion (standard deviation or interquartile range, respectively).

   Hypothesis contrast tests will be performed, with comparison of proportions when both variables are qualitative (Chi-square, Fisher's exact test) and comparisons of means for independent samples when one of them is quantitative (Student's t test if normal distribution or Mann-Whitney U test for variables that do not comply with normality). Survival will be estimated using the Kaplan-Meier method and survival curves will be compared using the Log-Rank test to analyze the effect of the different factors that may influence survival. The results of the study will be analyzed by intention-to-treat. After recruitment of half of the patients, an intermediate data analysis will be performed.

   The final analysis will be performed in two phases, one on the morbidity-mortality results at the end of recruitment, and another at the end of the study with the definitive data on recurrence and survival.

   A logistic regression model will be performed to evaluate the effect of representative covariates on the LRS. For this purpose, those that are significant in the univariate analysis (p<0.2) or clinically relevant will be included.

   A value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed primary gastric adenocarcinoma
* Clinical stages Ib, II and III of gastric cancer (8th edition of the TNM classification)
* Patients with ECOG Performance Status 0, 1 or 2
* Patients who sign the informed consent to participate in the study
* Patients over 18 years old
* Patients treated by surgery with curative intent
* Patients must be suitable for surgery.

Exclusion criteria:

* Any histology other than adenocarcinoma
* Stage Ia and IV
* Unresectability criteria (tumor factors): distant metastasis, peritoneal carcinomatosis, positive cytology of ascitic fluid, invasion or tumor entrapment of large vessels (aorta, liver, celiac trunk), infiltration of the root of the mesentery, para-aortic lymphadenopathy or levels >3, linitis plastica, involvement of other organs
* Inoperability criteria (patient factors): serious concomitant systemic disorders incompatible with surgery or the study (at the discretion of the investigator)
* Patients undergoing surgery for gastric cancer with open approach at the beginning
* Palliative surgery cases
* Non-compliance with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients with a diagnosis of gastric adenocarcinoma, histologically confirmed, whose preoperative extension study is compatible with stages IB, II and III of the 8th edition of the TNM classification (AJCC), in whom there is an indication for surgical treatment with curative intent by minimally invasive gastrectomy (RAG or LG), with or without neoadjuvant treatment, will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-13 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of clinical safety. | Intraoperative and Postoperative (up to 90 days postoperative)
  Intraoperative blood loss and perioperative complications (types of complications, Clavien Dindo classification, Comprehensive Complication Index (CCI®))
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of oncologic safety. | Intraoperative
  Nodal count (number of lymph nodes retrieved) and R0 resection margin.

SECONDARY OUTCOMES:
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of intraoperative outcomes. | Intraoperative
  * Operative time (duration of the surgical procedure measured in minutes)
  * Number of surgeons who have participated in the operation (1 to 5)
  * Need for conversion to open surgery (conversion to open surgery vs non-conversion)
  * Comfort of the surgeon during the intervention, using an analog scale of 0-5 (0 is no comfort, 1 is little comfort, 2 is moderate comfort, 3 is quite a bit of comfort, 4 is a lot of comfort and 5 is extreme comfort)
  * Learning curve (number of robotic versus laparoscopic gastrectomies performed by the surgeon before the registered case)
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of recovery and postoperative physical status. | Postoperative, up to 1 year after surgery
  * Onset of oral tolerance (measured in number of days from the intervention to the first oral intake)
  * Onset of mobilization (measured in number of days from the operation to the start of the patient's ambulation)
  * Hospital stay (number of days of hospital admission, counted from the day of the intervention until discharge)
  * Readmission (yes /no) (need for hospital admission after discharge, related to the operation, over 1 year postoperatively)
  * Mortality (yes /no) (procedure-related death, within 1 year postoperatively) In case of death: time in days since surgery.
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of oncological outcomes. | Assessment at 1, 3, 5 years from surgery
  * Overall survival (OS): time between the date of intervention and the date of death (from any cause).
  * Recurrence-free survival (RFS): time from the date of intervention to locoregional recurrence, distant recurrence or death, whichever occurred first. The date of biopsy will be the date of recurrence (or date of death).
  * Local recurrence: surgical site of gastrectomy and lymphadenectomy (anastomosis or perianastomosis nodes).
  * Distant or systemic recurrence: extra-regional lymph nodes (N3 and/or more distant lymph node levels), metastases in laparoscopic ports, parenchymal organ, carcinomatosis or bone metastases.
Compare robotic gastrectomy with the conventional laparoscopic approach in terms of cost-utility outcomes. | Assessment at 1 year from surgery
  Quality Adjusted Life Year (QALY).

CONTACTS AND LOCATIONS:
Overall Officials: Mª Asunción Acosta Mérida, MD. PhD., Principal Investigator — Department of General and Digestive Surgery, Dr. Negrin University Hospital of Gran Canaria
Locations (1):
- Mª Asunción Acosta Mérida, Las Palmas de Gran Canaria, Las Palmas, Spain